CLINICAL TRIAL: NCT07023783
Title: Using a Transdiagnostic Sleep Health Intervention Approach to Improve Sleep Quality and Subsequent Daytime Fatigue, Physical Activity, and Quality of Life in Cancer Survivors
Brief Title: Improving Sleep, Fatigue, Activity & Quality of Life in Cancer Survivors Via a Transdiagnostic Intervention
Acronym: SLEEP-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 776250
Record Dates: First submitted 2025-05-29; First posted 2025-06-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cancer Survivors
Keywords: Sleep Health; Physical Activity; Cancer Related Fatigue
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Health Intervention Arm (Experimental): A transdiagnostic sleep health intervention (TSHI) will be delivered across six weekly 50-minute one-on-one sessions with a sleep expert via a HIPAA-compliant videoconference link. The six weekly TSHI sessions are outlined as:
  Week 1: Consists of discussing sleep physiology and discussing appropriate bed and wake up times.
  Week 2: Consists of discussing how to set/importance of setting, a bedtime routine Week 3: Consists of discussing how to improve daytime function through energy management for daily and weekly tasks.
  Week 4: Consists of discussing the sleep beliefs the participant holds and possible corrections of any unhelpful sleep beliefs.
  Week 5: Consists of educating participants on sleep hygiene and how it is influenced by environmental, social, and physical factors.
  Week 6: Consists of discussing sleep behavior changes observed during the TSHI and collaborating with the participant on plans to maintain their new sleep pattern.
  Interventions: Behavioral: Transdiagnostic Sleep Health Intervention (TSHI)

INTERVENTIONS:
Behavioral: Transdiagnostic Sleep Health Intervention (TSHI) — A transdiagnostic sleep health intervention (TSHI) will be delivered across six weekly 50-minute one-on-one sessions with a sleep expert via a HIPAA-compliant videoconference link. The six weekly TSHI sessions are outlined as:
  Week 1: Consists of discussing sleep physiology and discussing appropriate bed and wake up times.
  Week 2: Consists of discussing how to set/importance of setting, a bedtime routine Week 3: Consists of discussing how to improve daytime function through energy management for daily and weekly tasks.
  Week 4: Consists of discussing the sleep beliefs the participant holds and possible corrections of any unhelpful sleep beliefs.
  Week 5: Consists of educating participants on sleep hygiene and how it is influenced by environmental, social, and physical factors.
  Week 6: Consists of discussing sleep behavior changes observed during the TSHI and collaborating with the participant on plans to maintain their new sleep pattern.

SUMMARY:
Poor sleep affects over half of U.S. cancer survivors, contributing to daytime fatigue, reduced physical activity, and diminished quality of life. Traditional sleep treatments often target diagnosed disorders, leaving many survivors with subclinical sleep issues underserved. Sleep health-a broader concept encompassing sleep regularity, satisfaction, alertness, timing, efficiency, and duration (RU-SATED)-offers a more inclusive framework for intervention. The TSHI is a modular, skills-based program designed to improve these dimensions of sleep health. Delivered via six weekly one-on-one Zoom sessions, TSHI emphasizes behavioral strategies like sleep hygiene, relaxation, and energy management.

This six-week, single-group quasi-experimental pilot study will enroll 10 cancer survivors to assess the feasibility, acceptability, and preliminary effectiveness of TSHI. Researchers will evaluate changes in sleep health, fatigue, physical activity, and quality of life using surveys, interviews, and ActiGraph data. By targeting sleep as a modifiable health behavior, this study aims to lay the groundwork for scalable interventions that enhance recovery and well-being in cancer survivors.

DETAILED DESCRIPTION:
While cancer incidence remains steady, survivorship is rapidly increasing, with over 18 million cancer survivors (CS) in the U.S. as of 2022 and projections estimating 26 million by 2040. As survival rates improve, attention has shifted toward enhancing the quality of life (QoL) for survivors. One of the most prevalent and under-addressed issues affecting CS is poor sleep health. More than half of survivors report sleep disturbances, which can persist long after treatment ends and are linked to fatigue, reduced physical activity, and diminished health-related quality of life (HRQoL). Despite the high prevalence, many survivors do not meet diagnostic criteria for sleep disorders and are thus excluded from traditional interventions like cognitive behavioral therapy for insomnia (CBT-I).

Sleep health is increasingly recognized as a multidimensional construct encompassing regularity, satisfaction, alertness, timing, efficiency, and duration (RU-SATED). This broader framework allows for interventions that target sleep as a modifiable behavior rather than a binary clinical diagnosis. The Transdiagnostic Sleep Health Intervention (TSHI) was developed to address these six dimensions through a modular, skills-based approach. TSHI is designed to be flexible, accessible, and scalable-delivered via six weekly 50-minute one-on-one sessions with a sleep expert through a HIPAA-compliant Zoom platform.

TSHI incorporates evidence-based strategies such as stimulus control, sleep restriction, relaxation techniques, energy management, cognitive restructuring, and sleep hygiene education. Each session builds on the last, guiding participants through personalized behavior change strategies aimed at improving sleep health and, by extension, daytime functioning and overall well-being.

To evaluate the feasibility and preliminary efficacy of TSHI in cancer survivors, the investigators are conducting a six-week, single-group, quasi-experimental pilot study with 10 participants. The study will assess both the acceptability of the intervention and its impact on key outcomes including sleep health, fatigue, physical activity, and HRQoL.

Participants will first complete baseline assessments, including validated surveys and one week of continuous monitoring using ActiGraph accelerometers to capture objective sleep and activity data. They will then engage in the six-session TSHI program. Following the intervention, participants will repeat the surveys and ActiGraph monitoring, and participate in semi-structured interviews to provide qualitative feedback on their experience.

Our primary aim is to determine whether TSHI is feasible and acceptable when delivered virtually to cancer survivors. The investigators hypothesize that participants will report high usability and satisfaction, with at least 80% retention and adherence.

Our secondary aim is to explore changes in RU-SATED sleep health dimensions, fatigue, physical activity, and HRQoL from pre- to post-intervention. The investigators expect to observe improvements across these domains, supported by both self-report and objective data.

Quantitative data will be analyzed using descriptive statistics and pre-post comparisons, while qualitative data from interviews will be thematically coded to identify common experiences and suggestions for refinement. This mixed-methods approach will provide a comprehensive understanding of TSHI's potential and inform future, larger-scale trials.

This project represents a critical step toward addressing the unmet sleep health needs of cancer survivors. By targeting sleep as a modifiable behavior and using a transdiagnostic framework, TSHI offers a promising, scalable solution to improve survivorship outcomes and enhance long-term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* ≤7 on RU-SATED questionnaire
* ≥6 months removed from primary cancer treatment
* able to speak/read English
* can sign informed consent
* have internet access via smartphone or computer

Exclusion Criteria:

* ≥15 on Patent Health Questionnaire 8
* ≥10 on Generalized Anxiety Disorder-7
* self-reported current or recent history (≤2 years) of drug or alcohol abuse
* history of nervous system disorder [e.g., stroke, Parkinson's disease, multiple sclerosis]
* severe mental illness such as schizophrenia or bipolar disorder
* current or recent history (≤5 years) of shift work
* currently receiving a sleep intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of a videoconference-based Transdiagnostic Sleep Health Intervention | After study week 7
  TSHI acceptability will be assessed qualitatively and quantitatively following the study. Qualitative assessments will involve semi-structured interviews with each participant, guided by a written list of questions. Quantitative assessments of TSHI acceptability, usability, and usefulness will use a modified System Usability Scale (SUS). scores range from 0-100 with a higher score indicating better perceived usability of the intervention.
Recruitment | After study week 7
  The investigators will assess program feasibility via recruitment. Recruitment rates will be: # of cancer survivors enrolled ÷ # of cancer survivors who complete the screening survey. With a higher number indicating ease, practicality, and efficiency of the recruitment process.
Study Retention | After study week 7
  We will assess program feasibility via study retention. Study retention will be: # of cancer survivors completing the TSHI ÷ # of cancer survivors who began the TSHI. A high retention rate indicates the ability to keep participants committed over time, suggesting that the project is feasible and likely to succeed.
Adherence Rates | After study week 7
  We will assess program feasibility via protocol adherence rates. Adherence will be: # of weekly videoconference-based TSHI sessions attended ÷ six (total number of TSHI sessions). A high adherence rate indicates that the study design is viable and participants are able and willing to follow the protocol.

SECONDARY OUTCOMES:
Changes in Sleep Health constructs | Baseline and After study week 6
  Means and standard deviations will be calculated to evaluate the pre/post difference in the Regularity, Satisfaction, Alertness, Timing, Efficiency, and duration sleep health scale ( RU-SATED constructs). During the Baseline and Post-Study Testing Sessions, participants will complete the RU-SATED scale. This validated six-item scale assesses sleep regularity, satisfaction, alertness, timing, efficiency, and duration (i.e., RU-SATED). A scores range from 0-12 with a higher score indicating healthier sleep health.
Sleep Regularity | Baseline and After Study week 6
  We will supplement RU-SATED construct measurements with sleep measurements made via the ActiGraph. Using the ActiGraph, Regularity will be assessed by the standard deviation of sleep midpoint, which is calculated as [sleep onset+(wake-sleep inset/2)]. The cut off for good sleep health is <60 minutes
Sleep Satisfaction | Baseline and After Study week 6
  Using the sleep log, satisfaction will be assessed. The sleep log includes an item to rate "restedness upon awakening" with 0= " not at all", 1 "somewhat"., 2= "moderately", 3= " quite a bit", and 4 = " extremely". Satisfaction will be operationalized as the average "restedness" score. the cut off for good sleep ehalth is an average of ≥3
Alertness | Baseline and After Study week 6
  Using the Epworth Sleepiness Scale, Alertness will be measured. The Epworth Sleepiness Scale consists of 8-items of various activities (ie. Sitting and reading, watching TV, etc) answered using a 4-point Likert scale with 0+ " would never nod off" to 3= "high chance of nodding off". The cut off for food sleep health is ≤ 10.
Timeing | Baseline and After Study week 6
  Using Actigraphy timing will be assessed. The Actigraphy measure of the average sleep midpoint will be used. The cut off for good sleep health is 2-4 AM.
Sleep Effiency | Baseline and After Study week 6
  To measure Efficiency Actigraphy will be used. The average total minutes of sleep divided by the time in bed multiplied by 100. A higher percentage indicates high sleep efficiency. The cut off for good sleep health is ≥ 85%
Sleep Duration | Baseline and After Study week 6
  To measure Duration Actigraphy will be used based on the average total minutes of sleep. the cut off for good sleep health is 6-8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma College of Allied Health, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No